CLINICAL TRIAL: NCT01764061
Title: Clinical Investigational Protocol for 2 RBC Single Unit Recovery on MCS®+ 8150 Using LN832 Disposable Sets (US)
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100067
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Red Blood Cell Donation
Keywords: Red Cells; Blood donors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to validate that single units of RBCs collected by the Haemonetics MCS®+ 8150 system using LN832 disposable sets during an interrupted double red cell collection protocol meet all in vitro FDA requirements for non-leukoreduced red blood cells, and to provide data to support the 510(k) clearance of the MCS®+ 8150 system using LN832 disposable sets for this intended use.

DETAILED DESCRIPTION:
This study will take place at two sites (Blood Center of Wisconsin (BCW) Milwaukee, WI and American Red Cross-Norfolk, VA).

* A standard double red cell collection protocol will be initiated using the Haemonetics MCS®+ 8150 system using LN832 disposable sets. The collection procedure will be terminated after collection of one RBC unit. The maximum target red cell volume will be selected based on the donor predonation weight as specified in the nomogram included in the MCS®+ 8150 operation manual.
* The RBC units will be stored for 42 days at 1° to 6°C.
* Upon collection and at 42 days after collection, the RBC units will be weighed and tested for hematology parameters (white blood cell count, red blood cell count, residual white blood cell count, hemoglobin, hematocrit, platelet count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red blood cell distribution width, and supernatant hemoglobin) and chemistry parameters (pH, potassium, glucose, lactate, and ATP).
* Acceptance criteria for this study are as follows:

  1. Hemolysis of less than or equal to 1% at 42 days of storage
  2. Maximum absolute red cell volume is less than or equal to the programmed absolute RBC target volume + 15%
  3. Minimum absolute red cell volume is greater than or equal to the programmed absolute RBC target volume - 15%
* After collection of sixty (60) evaluable RBC units, the study will be considered supportive of the intended use noted above if zero (0) units fail the acceptance criteria.
* If one (1) unit fails acceptance criteria after collection of sixty (60) evaluable RBC units, an additional seventy one (71) units will be collected.
* The study will be considered supportive of the intended use noted above if not more than one (1) total unit out of 131 evaluable units fails the acceptance criteria.
* If a total of two (2) units fail acceptance criteria, the study will not be considered supportive of the intended use noted above.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ≥ 18 years of age
* Males ≥ 130 pounds, Females ≥ 150 pounds
* Males ≥ 5 feet, 1 inch, Females ≥ 5 feet, 3 inches
* Hemoglobin ≥ 13.3 g/dL
* Hematocrit ≥ 40%
* Donor Eligibility: Meets all criteria as per sites' Research Blood Donation Record, Prior donation date (i.e. not less than 112 days for most recent double RBC unit donation, 56 days for most recent single RBC unit donation)
* Subject must provide informed consent using an IRB informed consent form prior to undergoing any study related procedures.

Exclusion Criteria:

* will be not fulfilling any of the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy blood donors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hemolysis level at 42 days of storage | 42 days
Absolute red cell volume | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Lou Anne Young Maes, MD, Principal Investigator — American National Red Cross; Jerome Gottschall, MD, Principal Investigator — Versiti Blood Health
Locations (2):
- United States (2):
  - American Red Cross, Norfolk, Virginia
  - Blood Center of Wisconsin, Milwaukee, Wisconsin